CLINICAL TRIAL: NCT01988662
Title: A 3 Months, patient-and Rater Blinded, Randomized, Prospective Study Comparing Systemic Anti-VEGF Effects Between Ranibizumab and Aflibercept in Treatment naïve Neovascular Age-related Macular Degeneration (nAMD) Patients
Brief Title: UNcovering the Difference Between Ranibizumab and Aflibercept, Focusing on Systemic Anti-vascular Endothelial Growth Factor (VEGF) Effects in Patients With neovascuLar Age-related Macular Degeneration (AMD)
Acronym: UNRAVEL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRFB002A-MAX-IL-01; 2013-003482-34 (EudraCT Number)
Record Dates: First submitted 2013-11-14; First posted 2013-11-20 (Estimated); Results first posted 2017-02-28 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-03

CONDITIONS: Neovacular Age-related Macular Degeneration
Keywords: nAMD, VEGF, VEGF agent, BCVA, CRT, Ranibizumab, Lucentis, Aflibercept, Eylea
MeSH Terms: conditions — Creatine deficiency, X-linked | interventions — Ranibizumab; aflibercept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranibizumab (Experimental): 104 patients with an eligible study eye were randomized to be treated with Ranibizumab IVT. 0.5 mg of commercially available Ranibizumab were used for intravitreal injection adminstered by an unblinded injecting physician. 3 injections were performed (Baseline, Month 1, Month 2).
  Interventions: Procedure: Neovascular Age-related Macular Degeneration
- Aflibercept (Active Comparator): 101 patients with an eligible study eye were randomized to be treated with Aflibercept IVT. 2.0 mg of commercially available Aflibercept were used for intravitreal injection admistered by an unblinded injecting physician. 3 injections were performed (Baseline, Month 1, Month 2).
  Interventions: Procedure: Neovascular Age-related Macular Degeneration

INTERVENTIONS:
Procedure: Neovascular Age-related Macular Degeneration — Blood measurement
  Other Names: Lucentis, Eylea

SUMMARY:
This study assessed systemic vascular endothelial growth factor (VEGF) level in patients with neovascular Age-related Macular Degeneration following treatment with Ranibizumab or Aflibercept.

Free plasma VEGF-A level was measured in this study .

ELIGIBILITY:
Key Inclusion Criteria

* Newly diagnosed Age-related Macular Degeneration (AMD)
* No previous treatment received for diagnosed AMD
* Visual Acuity 6/7.5 to 6/96

Key Exclusion Criteria:

* standard exclusion criteria for anti-VEGF treatment
* Visual Acuity <6/96
* nAMD in both eyes, or any condition in other eye which may have required anti- VEGF treatment during study period
* other disease in candidate eye which could have compromised visual acuity or required medical/surgical intervention during study period
* participation to other clinical study with 'not approved' treatment within a year prior to UNRAVEL study participation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2014-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (20):
- Israel (6):
  - Novartis Investigative Site, Beersheba
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Rehovot
  - Novartis Investigative Site, Tel Aviv
- Malaysia (2):
  - Novartis Investigative Site, Petaling Jaya, Selangor
  - Novartis Investigative Site, Kuala Lumpur
- Philippines (3):
  - Novartis Investigative Site, Makati City
  - Novartis Investigative Site, Pasig
  - Novartis Investigative Site, Quezon City
- Singapore (2):
  - Novartis Investigative Site, Singapore, Singapore
  - Novartis Investigative Site, Singapore
- South Korea (3):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Seoul
- Taiwan (2):
  - Novartis Investigative Site, Taipei, Taiwan
  - Novartis Investigative Site, Linkou District
- Thailand (2):
  - Novartis Investigative Site, Bangkok, Bangkoknoi
  - Novartis Investigative Site, Bangkok

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All randomized patients were included in the Full Analysis Set (FAS).
Groups:
- Ranibizumab: 104 patients with an eligible study eye were randomized to be treated with Ranibizumab IVT. 0.5 mg of commercially available Ranibizumab were used for intravitreal injection administered by an unblinded injecting physician. 3 injections were performed (Baseline, Month 1, Month 2).
- Aflibercept: 101 patients with an eligible study eye were randomized to be treated with Aflibercept IVT. 2.0 mg of commercially available Aflibercept were used for intravitreal injection administered by an unblinded injecting physician. 3 injections were performed (Baseline, Month 1, Month 2).
Period: Overall Study
Arm/Group | Ranibizumab | Aflibercept
Started | 104 | 101
Completed | 100 | 99
Not Completed | 4 | 2
Not completed — Subject/guardian decision | 1 | 1
Not completed — Adverse Event | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranibizumab | Aflibercept | Total
Number analyzed (Participants) | 104 | 101 | 205
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.1 (9.00) | 72.0 (8.43) | 71.0 (8.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 44 | 86
  Male | 62 | 57 | 119

OUTCOME MEASURES:

1. Secondary Outcome: Percent Change From Baseline in Plasma VEGF Level Overtime
Description: Plasma VEGF measurement performed at all visits and compared to baseline level
Time Frame: Change from baseline up to month 3
Population: FAS: The FAS consisted of all randomized patients who received at least one dose of study treatment. FAS was the analysis set. However, patients who were randomized due to erroneous use of the IRT system and who did not receive at least one dose of study treatment were excluded from the FAS.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Ranibizumab | Aflibercept
Number analyzed (Participants) | 104 | 101
Percent change
  Baseline (post-IVT injection; n=104, 100) | 11.93 (5.836) | -9.37 (6.100)
  Week 1 (n=103, 101) | 44.08 (14.377) | -7.44 (14.722)
  Week 2 (n=102, 100) | 38.76 (11.165) | -16.45 (11.434)
  Month 1 (pre-IVT injection; n= 102, 100)) | 112.05 (60.182) | 23.12 (61.641)
  Month 1 (post-IVT injection; n=101, 100) | 12.27 (6.711) | -20.61 (6.861)
  Month 2 (pre-IVT injection; n=100, 99) | 10.78 (7.342) | -19.13 (7.519)
  Month 2 (post-IVT injection; n=100, 99) | 50.59 (19.076) | -16.09 (19.535)
  Month 3 (n=100, 99) | 41.04 (19.918) | -21.53 (20.398)

2. Secondary Outcome: Correlation Between Percent Change From Baseline Plasma VEGF Level and the Serum Anti-VEGF Agent Overtime
Description: VEGF level and anti-VEGF concentration measured in the blood at each single visit, including pre- and post-dose measurement at the dosing visits.
Time Frame: pre-dose to post-dose at Baseline, week 1, week 2, month 1, month 2, and month 3
Population: FAS
Measure: Number (95% Confidence Interval); unit: pearson correlation coefficient
Arm/Group | Ranibizumab | Aflibercept
Number analyzed (Participants) | 104 | 101
pearson correlation coefficient
  Baseline (post-IVT injection) | -0.141 [-0.34 to 0.07] | 0.083 [-0.12 to 0.28]
  Week 1 | 0.027 [-0.17 to 0.22] | 0.234 [0.04 to 0.41]
  Week 2 | -0.085 [-0.28 to 0.11] | 0.192 [-0.01 to 0.37]
  Month 1 (pre-IVT injection) | -0.065 [-0.26 to 0.13] | 0.127 [-0.07 to 0.32]
  Month 1 (post-IVT injection) | -0.110 [-0.30 to 0.09] | 0.088 [-0.11 to 0.28]
  Month 2 (pre-IVT injection) | -0.151 [-0.34 to 0.05] | 0.051 [-0.15 to 0.25]
  Month 2 (post-IVT injection) | -0.049 [-0.25 to 0.15] | 0.098 [-0.10 to 0.29]
  Month 3 | -0.047 [-0.24 to 0.15] | 0.229 [0.03 to 0.41]

3. Secondary Outcome: Mean Change From Baseline in Best Corrected Visual Acuity (BCVA) of the Study Eye Over Time
Description: BCVA score is assessed on study eye based on the number of letters read correctly on the Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity charts at a testing distance of 4 meters. An increase in score indicates an improvement in acuity. Change from baseline calculated as observed post-baseline value - baseline value.
Time Frame: Baseline, month 1, month 2, month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Letter
Arm/Group | Ranibizumab | Aflibercept
Number analyzed (Participants) | 104 | 101
Letter
  Change at month 1 (n= 99, 100) | 3.9 (7.45) | 2.8 (9.7)
  Change at month 2 (n=98, 99) | 5.8 (8.54) | 5.1 (9.72)
  Change at month 3 (n= 99, 99) | 6.1 (8.36) | 6.9 (11.68)

4. Secondary Outcome: Mean Change From Baseline in Central Retinal Thickness (CRT) of the Study Eye Over Time
Description: CRT in micrometers assessed by Optical Tomography (OCT) at each single study visit. A reduction is thickness indicates an improvement is the lesion area.
  Change from baseline calculated as observed post-baseline - baseline value.
Time Frame: Baseline, month 1, month 2, month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Ranibizumab | Aflibercept
Number analyzed (Participants) | 104 | 101
micrometers
  Change at month 1 (n= 101, 100) | -75.0 (91.04) | -93.8 (106.43)
  Change at month 2 (n= 100, 99) | -94.3 (103.41) | -116.6 (123.35)
  Change at month 3 (n= 100, 99) | -93.7 (110.41) | -124.3 (122.46)

5. Secondary Outcome: Number of Patients With Ocular and Systemic Adverse Events
Description: The incidence of reported treatment emergent adverse events (TEAEs) and treatment emergent serious adverse events (TESAE).
Time Frame: Day 1 to day 85
Population: Safety (SAF) analysis set: The SAF analysis set included all patients who received at least one dose of study treatment and had at least one post-baseline safety assessment.
Measure: Number; unit: Participants
Arm/Group | Ranibizumab | Aflibercept
Number analyzed (Participants) | 104 | 101
Participants
  TEAEs | 32 | 32
  TESAEs | 3 | 5
  TEAEs leading to death | 0 | 0
  TEAEs with suspected relationship to study drug | 6 | 4
  TESAEs with suspected relationship to study drug | 1 | 0
  TEAEs w/ suspected relationship to ocular inject. | 12 | 11
  TESAEs w/ suspected relationship to ocular inject. | 1 | 0
  TEAEs leading to disc. of study treatment | 3 | 1

6. Primary Outcome: Percent Change From Baseline at Month 3 in Plasma VEGF Following Intravitreal (IVT) Injection of Anti-VEGF Agent
Description: Percent change in blood VEGF level is calculated as the difference in blood VEGF level measured after 3 month of anti-VEGF agent IVT treatment (Ranibizumab or Aflibercept) when compared to baseline blood VEGF level.
Time Frame: Change from baseline at Month 3
Population: Full Analysis Set (FAS): The FAS consisted of all randomized patients who received at least one dose of study treatment. FAS was the analysis set. However, patients who were randomized due to erroneous use of the IRT system and who did not receive at least one dose of study treatment were excluded from the FAS.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Ranibizumab | Aflibercept
Number analyzed (Participants) | 100 | 99
Percent change | 41.04 (19.918) | -21.53 (20.398)
Statistical Analysis 1: Comparison: Ranibizumab vs Aflibercept; H0: μR = μA versus HA: μR ≠ μA; Test type: Non-Inferiority or Equivalence — H0: There is no difference in the percent change in VEGF level after 3 months for patients with nAMD treated with ranibizumab compared to aflibercept. HA: There is a difference in the percent change in VEGF level after 3 months for patients with nAMD treated with ranibizumab compared to aflibercept; p = 0.012, Mixed Models Analysis; Mean Difference (Net) = 62.57, 95% CI 2-sided [13.96 to 111.17], Standard Error of Mean 24.639

ADVERSE EVENTS:
Time Frame: Throughout the study period (day 1 to day 85)
Description: Safety assessments consisted of collecting all AEs, serious adverse events (SAEs), with their severity and relationship to study drug and ocular injection, and pregnancies.
Arm/Group | Ranibizumab | Aflibercept | Total
Serious Adverse Events (participants affected / at risk) | 3/104 | 5/101 | 8/205
Other Adverse Events (participants affected / at risk) | 20/104 | 19/101 | 39/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab (N=104) | Aflibercept (N=101) | Total (N=205)
Retinal haemorrhage (Eye disorders) | 1 | 1 | 2
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab (N=104) | Aflibercept (N=101) | Total (N=205)
Conjunctival haemorrhage (Eye disorders) | 8 | 8 | 16
Conjunctival hyperaemia (Eye disorders) | 2 | 1 | 3
Dry eye (Eye disorders) | 3 | 1 | 4
Eye inflammation (Eye disorders) | 2 | 0 | 2
Eye pain (Eye disorders) | 4 | 3 | 7
Punctate keratitis (Eye disorders) | 3 | 2 | 5
Visual acuity reduced (Eye disorders) | 2 | 2 | 4
Vitreous floaters (Eye disorders) | 2 | 2 | 4
Sensation of foreign body (General disorders) | 3 | 1 | 4
Nasopharyngitis (Infections and infestations) | 1 | 2 | 3
Blood pressure increased (Investigations) | 2 | 2 | 4
Intraocular pressure increased (Investigations) | 0 | 2 | 2
Dizziness (Nervous system disorders) | 0 | 2 | 2
Headache (Nervous system disorders) | 3 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigators from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.